CLINICAL TRIAL: NCT06438198
Title: Unraveling the (patho)physiological Mechanisms and Potential Clinical Benefits of an Early Switch from Controlled to Assisted Ventilation
Brief Title: Early Switch from Controlled to Assisted Ventilation
Acronym: SWITCH-SAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Annemijn Jonkman, Assistant Professor, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MEC-2024-0011
Record Dates: First submitted 2024-05-14; First posted 2024-05-31 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Acute Hypoxemic Respiratory Failure; Mechanical Ventilation
Keywords: Electrical Impedance Tomography; Esophageal manometry; Controlled Mechanical Ventilation; Assisted Mechanical Ventilation; Respiratory Monitoring
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mechanically ventilated adults (Experimental): Switch from controlled to assisted mechanical ventilation when PaO2/FiO2-ratio > 200 mmHg.
  Before switch (on controlled ventilation) participants will undergo an electrical impedance tomography (EIT) perfusion measurement as well as a photon-counting CT (PCCT) scan to assess lung perfusion and ventilation/perfusion mismatch. From 15 minutes before until 4 hours after switch and 30 minutes twice daily for 72 hours or until switch failure participants will be monitored continuously using EIT, esophageal pressure and gastric pressure.
  Interventions: Other: Pre-specified switch from controlled to assisted ventilation when PaO2/FiO2-ratio > 200 mmHg

INTERVENTIONS:
Other: Pre-specified switch from controlled to assisted ventilation when PaO2/FiO2-ratio > 200 mmHg — A pre-specified switch from controlled to assisted ventilation will be initiated when PaO2/FiO2-ratio > 200 mmHg. The moment of switch is pre-specified but patient management and ventilator settings are up to the clinical team. Switch is complete when the patient triggers all breaths spontaneously. Switch success is defined if patient reaches 72 hours on assisted ventilation. Switch failure is defined if patient switches back to controlled ventilation for more than 2 hours before 72 hours.

SUMMARY:
The goal of this physiological intervention study is to unravel the (patho)physiological mechanisms and potential clinical benefits of a pre-specified early switch from controlled to assisted ventilation in mechanically ventilated adult patients with acute hypoxemic respiratory failure (PaO2/FiO2 ratio < 200 mmHg).

The intervention is that participants will be switched from controlled to assisted ventilation when PaO2/FiO2 ratio > 200 mmHg.

The primary endpoint is the change in regional lung stress (as derived by electrical impedance tomography) when switching from controlled to assisted ventilation and until a successful or failed switch.

DETAILED DESCRIPTION:
A crucial milestone in the trajectory of the mechanically ventilated patient is the switch from fully controlled mechanical ventilation to assisted ventilation. This switch should be made as early as feasible and safe, to limit the detrimental effects from prolonged controlled ventilation and sedation. However, there is also indirect evidence that excessive breathing effort during assisted ventilation may worsen lung injury (P-SILI). There are no guidelines that address this important switch moment.

Therefore, the overall aim of this physiological intervention study is to unravel the (patho)physiological mechanisms and potential clinical benefits of a pre-specified early switch from controlled to assisted ventilation in mechanically ventilated adult patients with acute hypoxemic respiratory failure (PaO2/FiO2 ratio < 200 mmHg).

Participants will be switched from controlled to assisted ventilation switch when PaO2/FiO2 ratio > 200 mmHg and will be monitored continuously using electrical impedance tomography, and oesophageal and gastric pressure until 4 hours post-switch and twice daily for 72 hours or until switch failure (switch back to controlled ventilation within 72 hours).

The primary endpoint is the change in regional lung stress (as derived by electrical impedance tomography) when switching from controlled to assisted ventilation and until a successful or failed switch.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Written informed consent from a legal representative
* Mechanical ventilation via an endotracheal tube
* Acute hypoxemic respiratory failure with PaO2/FiO2 ratio < 200 mmHg
* Under continuous sedation with or without paralysis

Exclusion Criteria:

* Expected mechanical ventilation duration of <48 hours
* Pure chronic obstructive pulmonary disease exacerbation
* Pre-existent respiratory muscle disease
* Contraindication to EIT monitoring (as per clinical protocol, e.g. pacemaker, burns or thoracic wounds limiting electrode placement)
* Contra-indications to oesophageal manometry (as per clinical protocol, e.g., recent oesophageal surgery, oesophageal varices, severe bleeding disorders)
* Known pregnancy
* Anticipating withdrawal of life support and/or shift to palliation as the goal of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Regional lung stress | 72 hours
  The change in regional lung stress as derived from EIT recordings by computing the regional ventilation distribution (ventral-to-dorsal ratio).

SECONDARY OUTCOMES:
Electrical Impedance Tomography (EIT) parameters | 72 hours
  Change in EIT parameters after transition from controlled to assisted ventilation (%)
Photon-Counting Computed Tomography (PCCT)-derived ventilation/perfusion mismatch | 30 minutes
  Ventilation/perfusion mismatch during controlled ventilation measured with photon-counting CT scan
Electrical Impedance Tomography (EIT)-derived ventilation/perfusion mismatch | 30 minutes
  Ventilation/perfusion mismatch during controlled ventilation measured with EIT
Respiratory mechanics | 72 hours
  Change in respiratory mechanics after transition from controlled to assisted ventilation (cmH2O)
Breathing effort | 72 hours
  Time-course of breathing effort during assisted ventilation as measured with esophageal manometry (cmH2O).
Patient-ventilator asynchrony | 72 hours
  Percentage of asynchronous breaths during assisted ventilation
Gas exchange | 72 hours
  Change in gas exchange after transition from controlled to assisted ventilation (%)
Hemodynamics | 72 hours
  Change in hemodynamics after transition from controlled to assisted ventilation (%)
Blood inflammatory biomarkers | 72 hours
  Blood biomarkers concentrations including cytokines and chemokines (i.e., interleukins, TNF-alpha, MCP-1 and MIP-1beta, CD14) measured as the difference between baseline vs. 72h (%)
Breath condensate inflammatory biomarkers | 72 hours
  Swivel-derived exhaled-breath condensate biomarkers concentrations including cytokines and chemokines (i.e., interleukins, TNF-alpha, MCP-1 and MIP-1beta, CD14) measured as the difference between baseline vs. 72h (%)
Ventilator-free days | 28 days
  Ventilator-free days at day 28

CONTACTS AND LOCATIONS:
Overall Officials: Annemijn Jonkman, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No